CLINICAL TRIAL: NCT06456086
Title: Effect of Epstein-Barr Virus on Macrophage M2/M1 Migration and EphA2 Expression in Adverse Drug Reactions
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Tang Junting, Director, First Affiliated Hospital of Kunming Medical University
Other Study IDs: 2023L88
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Adverse Drug Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stevens-Johnson syndrome/toxic epidermal necrolysis
  Interventions: Biological: stimulation with EB virus
- healthy control group
  Interventions: Biological: stimulation with EB virus
- Maculopapular Eruption
  Interventions: Biological: stimulation with EB virus

INTERVENTIONS:
Biological: stimulation with EB virus — stimulation with EB virus

SUMMARY:
This study aims to investigate the effect of EBV reactivation or EBV reactivation added with dexamethasone(DXM) in patients with adverse drug reactions(CDR) , through evaluating the levels on monocyte, macrophage M2/M1 and cytokines. To investigate whether expression of EBV receptors EphA2 could specifically influence on EBV activation in CDRs. We performed a prospective longitudinal study on the frequencies of Monocyte, Macrophage, M2/M1 and cytokines included IL-4,IL-13,TNF-α,IFN-γ,IFN-β, CXCL9 and CXCL10 after onset of MPE ,SJS/TEN and control groups. PBMCs collected from peripheral blood were cocultured with EBV or EBV with DXM. We next examined whether EBV or EBV with DXM could have a strong impact on the MOs, Mac, M2/M1 and cytokines and which cytokines could be crucial for the interaction between M2/M1 and EBV, by in vitro cocultures. Finally, EphA2 were detected to evaluate reactivation of EBV.

ELIGIBILITY:
Inclusion Criteria:

1. Age and Gender: The study includes male and female patients aged 18 years and older.
2. a.Erythema Multiforme (MPE) Patients: Diagnosed based on clinical presentation and medical examination findings.b.Stevens-Johnson Syndrome/Toxic Epidermal Necrolysis (SJS/TEN) Patients: Diagnosed according to the criteria set by the International Dermatology Society for SJS or TEN.c.Control Group: Healthy volunteers, without any history of chronic disease or acute infection, and not currently on any medications.

Exclusion Criteria:

1. Other Chronic Diseases: Patients with active heart, liver, kidney disease, or other systemic conditions.
2. Acute Infection: Patients who have had a viral or bacterial infection within the month prior to enrollment.
3. Immune Status: Patients who are immunocompromised or are receiving immunosuppressive therapy.
4. Allergy History: Patients with a known allergy to any drugs or agents used in the study.
5. Pregnancy or Lactation: Women who are currently pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Erythema Multiforme (MPE) Patients: Diagnosed based on clinical presentation and medical examination findings.or
  2. Stevens-Johnson Syndrome/Toxic Epidermal Necrolysis (SJS/TEN) Patients: Diagnosed according to the criteria set by the International Dermatology Society for SJS or TEN.or
  3. Control Group: Healthy volunteers, without any history of chronic disease or acute infection, and not currently on any medications.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
changes in the levels of monocytes, macrophages, M2/M1 ratio, and cytokines | 24 hours and 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Tang Junting, Kunming, Yunnan, China